CLINICAL TRIAL: NCT06292507
Title: Comparative Effects of Myofascial Stretch and Contract-relax Technique on Tone and Function of Upper Limb in Children With Spastic Cerebral Palsy
Brief Title: Comparative Effects of Myofascial Stretch and Contract-relax in Children With Spastic cp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0734
Record Dates: First submitted 2023-12-26; First posted 2024-03-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Myofascial stretch; Contract-Relax; Upper Limb
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFFECTS OF MYOFASCIAL STRETCH (Experimental): This group will receive Myofascial stretch Group.
  Interventions: Other: MYOFASCIAL STRETCH
- CONTRACT-RELAX TECHNIQUE ON TONE (Experimental): This group will receive Contract-Relax technique Group
  Interventions: Other: CONTRACT-RELAX TECHNIQUE

INTERVENTIONS:
Other: MYOFASCIAL STRETCH — Group A 10 participants will receive Myofascial Stretching
  Arms: EFFECTS OF MYOFASCIAL STRETCH
Other: CONTRACT-RELAX TECHNIQUE — group B 10 participants will receive Control-Relax Stretching Technique.
  Arms: CONTRACT-RELAX TECHNIQUE ON TONE

SUMMARY:
Cerebral palsy (CP) is primarily a neuromotor disorder that affects the development of movement, muscle tone and posture.It is one of the three most common lifelong developmental disabilities, the other two being autism and mental retardation causing considerable hardship to affected individuals and their families. CP is a common problem, the worldwide incidence being 2 to 2.5 per 1000 live births. Myofascial therapy is definable by "the facilitation of mechanical, neural and psycho physiological adaptive potential as interfaced by the myofascial system". The PNF contract-relax technique consists of stretching the target muscle, keeping it in position while the patient isometrically contracts it and relaxes in sequence, producing effects such as maintenance and gain in joint mobility, increased muscle strength, and better motor control whereas The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone This study will be randomized clinical trial and will be conducted in Rasool medical centre Gujrat and City hospital Gujrat. This study will be completed within duration of 6 months after the approval of synopsis.Convenience sampling technique will be used to collect the data. A sample size of total 20 patientswill be taken in the study. 20participants will be equally divided into two group's myofascial stretch and contract-relax stretching techniques having 10participants in each group. Informed consent will be sought from them and they will be clearly explained about the purpose of study.Myofascial Stretching will be applied to Group A and Contract-Relax stretching will be applied to Group B.

Results will be analyzed on SPSS.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is primarily a neuromotor disorder that affects the development of movement, muscle tone and posture. The underlying pathophysiology is an injury to the developing brain in the prenatal through neonatal period. Although the initial neuropathologic lesion is non-progressive, children with CP may develop a range of secondary conditions over time that will variably affect their functional abilities.

Cerebral palsy refers to set of lifelong mobility issues and postural defects which restrict function caused by non-progressive abnormalities in growing foetus or neonatal brain. CP is frequently followed by sensory, cognitive, behavioural impairment and musculoskeletal difficulties. CP could categorised as spastic, athetoid, ataxic, or mixed, also classed as hemiplegia, diplegia, quadriplegia, depending on kind of mobility dysfunction. Spasticity of numerous muscle groups is common in CP due to CNS injury

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 12 year(20).
* Spastic CP child will be including.
* Communication statusand oriented.
* Informed written consent of the children's parents was required.

Exclusion Criteria:

* Orthopedic surgery on upper limb(1).
* Received botulinum toxin injection in the upper limb during the last 6 months or who wish to receive it within the period of study(2).
* Upper Extremities deformities
* Upper limb Contracture Formation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Manual Ability Classification system | 4 month
  Psychometric properties of the MACS have been assessed with analysis of content, criterion, construct validity, and reliability. The intraclass correlation coefficient between therapists was 0.97 (95% confidence interval 0.96-0.98), and between parents and therapist was 0.96 (0.89-0.98), indicating excellent agreement

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Muhammad Farooq, MS*, Principal Investigator — Riphah International University
Locations (1):
- Mirza Muhammad Farooq, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choudhary A, Gulati S, Kabra M, Singh UP, Sankhyan N, Pandey RM, Kalra V. Efficacy of modified constraint induced movement therapy in improving upper limb function in children with hemiplegic cerebral palsy: a randomized controlled trial. Brain Dev. 2013 Oct;35(9):870-6. doi: 10.1016/j.braindev.2012.11.001. Epub 2012 Dec 11. PMID 23238223